CLINICAL TRIAL: NCT03041844
Title: Enhanced Ultrasound Treatment of Chronic Wounds With Monitoring of Healing and Quality of Life Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Drexel University (Other)
Collaborators: University of Pennsylvania (Other); Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1609004864
Record Dates: First submitted 2017-01-25; First posted 2017-02-03 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Foot Ulcer; Venous Ulcer
Keywords: therapeutic ultrasound; quality of life
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Frequency, Low Intensity Ultrasound (Experimental): Low Frequency, Low Intensity therapeutic ultrasound applied weekly for up to 16 weeks.
  Interventions: Device: Low Frequency, Low Intensity Ultrasound
- Sham Ultrasound (Sham Comparator): Sham ultrasound applied weekly for up to 16 weeks.
  Interventions: Device: Sham Applicator

INTERVENTIONS:
Device: Low Frequency, Low Intensity Ultrasound — Therapeutic ultrasound (20 kHz, <100 mW/cm2 spatial peak-temporal peak)
  Arms: Low Frequency, Low Intensity Ultrasound
Device: Sham Applicator — Sham ultrasound applicator
  Arms: Sham Ultrasound

SUMMARY:
The purpose of this study is to evaluate the effect of low frequency, low intensity ultrasound treatment on wound healing and health-related quality of life with a randomized clinical trial of patients with venous ulcers or diabetic ulcers.

DETAILED DESCRIPTION:
The two most common types of chronic wounds are venous ulcers (VUs) and diabetic ulcers (DUs). The investigators will conduct the first double-blind randomized controlled trial (RCT) to test the effect of low-frequency, low-intensity (LFLI) ultrasound (US) on chronic wound healing and health related quality of life (HRQOL) with high statistical confidence (α < 0.05, power > 0.90, n=60 VUs, n=60 DUs). The investigators' approach combines this active therapy with non-invasive diagnostic monitoring of wound hemodynamics throughout the treatment cycle, and includes analysis of the impact of nutritional status and inflammation on wound closure. There are several innovative aspects of this work. Specifically, (1) The lightweight, battery-powered applicator is the first potentially wearable ultrasound wound therapy device that is safe to apply for extended periods of time. (2) The applicator actively promotes healing, which is fundamentally different from commercial ultrasonic systems that remove necrotic tissue only. (3) The study approach will link LFLI US exposure to changes in wound hemodynamics and HRQOL, which has the potential to enable personalized medicine. (4) The analysis of patient nutritional and systemic inflammatory status may enable further treatment customization by identifying those patients most likely to benefit from LFLI US therapy. (5) The study approach incorporates both disease-specific and generic measures of HRQOL, which is unique for a therapeutic ultrasound RCT.

The low-frequency, low-intensity (20 kiloHertz (kHz), <100 milliWatt per square centimeter (mW/cm2) spatial peak-temporal peak), portable ultrasound applicator is lightweight (<25g) and permits safe and clinically pragmatic wound treatment. The field parameters of the US device were previously optimized for venous ulcers, and three recent pilot clinical human studies (VUs: n=20, n=25; DUs: n=10) demonstrated that the treatment improved healing by 15% per week compared to sham treatment. The investigators therefore anticipate that our treatment will accelerate closure of chronic wounds, and hypothesize that (1) LFLI US will improve generic and disease-specific HRQOL scores, (2) LFLI US will activate beneficial changes in the microvasculature of the wound and surrounding tissue, and (3) individuals with poor nutrition and high levels of inflammation will have delayed wound healing.

The specific aims are to: (1) Assess the effect of LFLI US on VUs and DUs by measuring wound closure as a primary endpoint and generic and disease-specific HRQOL as secondary endpoints. (2) Monitor the effects of LFLI US on wound perfusion and oxygenation using non-invasive optical methods, and (3) Determine the impact of nutritional status and inflammation on closure of DUs and VUs. Overall, this work will validate LFLI US as a safe, portable, and cost-effective therapy for chronic wounds. This is important because new therapies and improved clinical paradigms for wound management are urgently needed. Over the long-term, the study findings may enable the development of personalized wound treatment regimens across care settings.

ELIGIBILITY:
Inclusion Criteria:

* Have a venous ulcer (VU) or diabetic ulcer (DU) that has been documented for at least 8 weeks without complete re-epithelialization and is larger than 0.75 cm2 in size.
* VUs must be present on the lower extremities non-weight-bearing areas.
* DUs must be present on the ankle or foot and be secondary to complications from diabetes.
* Patients with DUs must have a documented history of diabetes mellitus of at least six months.

Exclusion Criteria:

* VUs secondary to any connective tissue disorder or blood dyscrasias.
* Severe vascular insufficiency (ankle-brachial index lower than 0.75 or toe-brachial index below 0.5).
* Active, untreated infection
* Acute deep venous thrombosis
* Cutaneous malignancy present on the involved extremity
* Active (or past 6 months) cancer treatment
* Presence of both a diabetic ulcer and a venous ulcer on the same extremity
* Known allergy to Tegaderm (a polyurethane dressing)
* Pregnant women
* Individuals younger than 18 years of age regardless of emancipation status
* Prisoners
* Individuals unable to speak English, Spanish, or Mandarin
* Adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01; Primary Completion 2022-03 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in wound size | 4 weeks
  Percentage change in wound size over 4 weeks

SECONDARY OUTCOMES:
Wound closure | 16 weeks
  Complete wound closure at 16 weeks
Health Related Quality of Life (HRQOL) | 16 weeks, then 6 and 12 months after last treatment
  Short form health survey will be administered to assess changes in HRQOL
Wound Quality of Life (WQOL) | 16 weeks
  Health survey will be administered to assess changes in wound-related HRQOL
Wound oxyhemoglobin concentration change | 16 weeks
  Change in wound oxyhemoglobin concentration per week, measured with diffuse near infrared spectroscopy (DNIRS)
Microcirculatory blood flow index change | 16 weeks
  Change in microcirculatory blood flow index per week, measured with diffuse correlation spectroscopy (DCS)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Lewin, PhD, Principal Investigator — Drexel University
Locations (1):
- Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided